CLINICAL TRIAL: NCT04634344
Title: A Phase I, Open-Label, Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics and Anti-tumor Efficacy of DZD2269 in Patients With Metastatic Castration Resistant Prostate Cancer
Brief Title: Assess the Safety, Tolerability, PK and Anti-tumor Efficacy of DZD2269 in Patients With MCRPC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to reasons of internal business strategy, not related to study or site conduct.
Sponsor: Dizal Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DZ2019A0001
Record Dates: First submitted 2020-11-02; First posted 2020-11-18 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Metastatic Castration Resistant Prostate Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DZD2269 as monotherapy (Experimental)
  Interventions: Drug: DZD2269

INTERVENTIONS:
Drug: DZD2269 — A single dose of DZD2269 starting at 5 mg will be given on Cycle 0 and then followed by a wash-out period. Multiple doses of DZD2269 at the same dose level will be given once daily after the wash-out period.

SUMMARY:
This study will treat patients with Metastatic Castration Resistant Prostate Cancer who have progressed following prior therapy. This is the first time this drug has ever been tested in patients, and so it will help to understand what type of side effects may occur with the drug treatment. It will also measure the the levels of drug in the body and preliminarily assess its anti-cancer activity as monotherapy.

DETAILED DESCRIPTION:
A first-time-in-human, Phase I, open-label, multicenter study to determine safety, tolerability, pharmacokinetics, and preliminary anti-tumor activity of DZD2269 in patients with mCRPC.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent form, taken prior to any study specific procedures, sampling and/or analyses.
2. Male patients age ≥ 18 years (≥ 19 in S. Korea), ECOG status 0-1, Predicted life expectancy ≥ 12 weeks,
3. All patients enrolled must have histologically confirmed diagnosis of adenocarcinoma of the prostate, with metastatic disease, and must also previously progressed on standard-of-care (SoC) therapy (i.e., abiraterone or enzalutamide, taxanes such as docetaxel or cabazitaxel) despite castrate levels of testosterone.
4. Be willing to provide blood samples and paired tumor tissue (if accessible) for the exploratory biomarker research
5. Total testosterone < 50 ng/dL at screening (except for subjects with prior orchiectomy, where testosterone does not need to be measured).
6. Adequate bone marrow reserve and organ system functions
7. LVEF ≥ 55% assessed by ECHO or MUGA

Exclusion Criteria:

1. Cytotoxic chemotherapy from a previous treatment regimen within 21 days of the first dose of study treatment.
2. Major surgery procedure (excluding placement of vascular access), or significant traumatic injury within 4 weeks of the first dose of study treatment, or have an anticipated need for major surgery during the study.
3. Prior exposure to therapeutic anticancer vaccines
4. Prior immune-mediated therapy including, but not be limited to, anti-CTLA-4, anti-PD1, anti-PDL1 and anti-PDL2 must have a wash-out period of ≥ 30 days before dosing
5. Prior/concomitant therapy with any other A2aR antagonist.
6. Live vaccines within 28 days prior to first dose.
7. Radiotherapy with a limited field for palliation within 1 week of the first dose of study treatment.
8. Patients currently receiving (or unable to stop using) medications or herbal supplements known to be potent inhibitors or inducers of CYP3A4, sensitive CYP3A4 substrates with narrow therapeutic index, and sensitive MATE1 and MATE2-K substrates with narrow therapeutic range
9. Any unresolved toxicities > Grade 1 (except alopecia).
10. Bone pain due to metastatic bone disease that cannot be managed with a routine, stable dose of a narcotic analgesic
11. Active infections as outlined in protocol
12. Spinal cord compression.
13. Patients who require systemic use of corticosteroids (at any dose)
14. Refractory nausea and vomiting if not controlled by supportive therapy
15. Cardiac criteria as outlined in protocol
16. Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer or other cancer from which the patient has been disease free for ≥ 2 years or which will not limit survival to < 2 years

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Incidence of AEs and SAEs | From screening to 28 days after the last dose
  To investigate the safety and tolerability of DZD2269 as monotherapy in patients with metastatic castration resistant prostate cancer (mCRPC)
Incidence of DLTs | From the first dose of study treatment up to the last day of Cycle 1 (28 days after start of multiple dosing)
  To establish Maximum Tolerated Dose (MTD) (if possible) in patients with mCRPC

SECONDARY OUTCOMES:
Drug concentrations of DZD2269 in plasma and urine | to approximately 6 months
  Pharmacokinetics endpoints
Maximum plasma concentration (Cmax) of DZD2269 | up to approximately 6 months
  Pharmacokinetics endpoints
Area under the plasma concentration-time curve (AUC) of DZD2269 | up to approximately 6 months
  Pharmacokinetics endpoints
Objective Response Rate (ORR) | Through the study completion, an average of around 1 year
  To assess the preliminary anti-tumor efficacy of DZD2269 as monotherapy based on modified RECIST
Disease Control Rate (DCR); | Through the study completion, an average of around 1 year
  To assess the preliminary anti-tumor efficacy of DZD2269 as monotherapy based on modified RECIST
Duration of Response (DoR) | Through the study completion, an average of around 1 year
  To assess the preliminary anti-tumor efficacy of DZD2269 as monotherapy based on modified RECIST

CONTACTS AND LOCATIONS:
Locations (6):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- South Korea (4):
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea - Seoul St. Marys Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bai Y, Zhang X, Zheng J, Liu Z, Yang Z, Zhang X. Overcoming high level adenosine-mediated immunosuppression by DZD2269, a potent and selective A2aR antagonist. J Exp Clin Cancer Res. 2022 Oct 14;41(1):302. doi: 10.1186/s13046-022-02511-1. PMID 36229853